CLINICAL TRIAL: NCT04430387
Title: Evaluation of Impact on Environmental Spatter Using Different Isolation Methods During Hygiene Appointment Among Pediatric Patients
Brief Title: Dental Isolation Methods in Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study initially aimed to measure droplets; however, as more was learned about COVID transmission, it became apparent that aerosol should be measured, but the method to measure aerosol was not possible for this study, so the study was withdrawn.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Di Wu, DDS MS PhD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-DB-20-0381
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Dental Plaque; Calculus, Dental; Aerosol Disease
Keywords: infection control; dental hygiene; spatter; aerosol
MeSH Terms: conditions — Dental Plaque; Dental Calculus

STUDY DESIGN:
Intervention Model Description: Recruited subjects will be randomly assigned to one of the three study groups for isolation during their dental cleaning, which are: Group 1- The saliva ejector; Group 2- The high-volume evacuator (HVE); Group 3- The DryShield.
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blind to group assignment of the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1- The saliva ejector (Active Comparator)
  Interventions: Device: The saliva ejector
- Group 2- The high-volume evacuator (Active Comparator)
  Interventions: Device: The high-volume evacuator
- Group 3- The DryShield (Active Comparator)
  Interventions: Device: The DryShield

INTERVENTIONS:
Device: The saliva ejector — A thin suction tube that draws water, saliva, blood, and debris from the mouth to provide patient comfort, preventing patient from constantly having to sit up and spit while maintain a clear operative field. It is connected through the low-volume suction hose in the dental chair. It can be held by the dental assistant, the dental provider or by the patient. In practice, it can be also contoured and hang by the cheek of the patient due to its light weight.
  Arms: Group 1- The saliva ejector
Device: The high-volume evacuator — The high-velocity air evacuation device. It is connected through the high-volume suction hose in the dental chair. It is operated by a dental assistant during the dental treatment, owing to the challenge posed by the rigid disposable attachment and bulky high-volume suction hose.
  Arms: Group 2- The high-volume evacuator
Device: The DryShield — The device is attached to the high-volume suction hose to provide continuous suction of intraoral fluid and debris, and also simultaneous isolation to both maxillary and mandibular quadrants on the same side. Other advantages of these devices include retracting the tongue and cheek, and prevention of aspiration.
  Arms: Group 3- The DryShield

SUMMARY:
The purpose of this study is to collect, measure, and assess the environmental spatter produced during dental appointments under different isolation methods used in pediatric dentistry, to compare the effectiveness of aerosol reduction between these methods, to identify the most effective way to manage aerosol during dental prophylaxis for pediatric patients and to provide clinical evidence to facilitate practice guidelines in dentistry related to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 patients
* Receiving dental prophylaxis or restorative procedure not requiring sedation or nitrous oxide
* Ability to cooperate in the dental chair
* Parents speak/read either English or Spanish and consent to study
* Child, when age appropriate, can assent to study

Exclusion Criteria:

* Patients that do not meet the above criteria (including inability to cooperate or special health care need)
* Parents that do not speak/read either English or Spanish
* Children that do not assent (when age appropriate) to the study

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
To collect, measure, and assess the environmental spatter produced during dental appointments under different isolation methods used in pediatric dentistry | Through case completion, an average a year
  The image of the spots of fluorescence from the spatter collected will be captured using a digital camera (Nikon D3100, Nikon, Tokyo, Japan) with an amber-colored lens cover. The image will be processed by a digital imaging software, ImageJ (National Institutes of Health, the Laboratory for Optical and Computational Instrumentation, University of Wisconsin) to get the number of the spots on each mask and film. The number of fluorescent spots is recorded to determine the amount of spatter produced.

CONTACTS AND LOCATIONS:
Overall Officials: Di I Wu, DDS,MS,PhD, Principal Investigator — UTHealth Science Center at Houston

IPD SHARING:
Plan to Share IPD: No
Not sharing

REFERENCES:
- [Derived] Kumbargere Nagraj S, Eachempati P, Paisi M, Nasser M, Sivaramakrishnan G, Verbeek JH. Interventions to reduce contaminated aerosols produced during dental procedures for preventing infectious diseases. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013686. doi: 10.1002/14651858.CD013686.pub2. PMID 33047816